CLINICAL TRIAL: NCT01779492
Title: A Randomized, Open-label, Multiple-dose, Two-sequence, Two-period Crossover Study to Investigate The Pharmacokinetics Between a GL2907 and Oxycontin CR Tab. 10mg in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GL Pharm Tech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GL2907-102
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: Oxycodone, controlled release formulation
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GL2907 (Experimental): Oxycodone HCl 20mg
  Interventions: Drug: GL2907
- Oxycontine CR 10mg (Active Comparator): Oxycodone HCl 10mg
  Interventions: Drug: Oxycontine CR 10mg

INTERVENTIONS:
Drug: GL2907 — once a day
  Other Names: Oxycodone HCl 20mg
  Arms: GL2907
Drug: Oxycontine CR 10mg — twice a day
  Other Names: Oxycodone HCl 10mg
  Arms: Oxycontine CR 10mg

SUMMARY:
The purpose of this clinical trial is to compare the pharmacokinetic characteristics of GL2907 XL 20mg tablet and Oxycontin CR 10mg tablet.

DETAILED DESCRIPTION:
GL2907 XL 20mg tablet is controlled released formulation which is made by GL Pharm Tech.

ELIGIBILITY:
Inclusion Criteria:

* 20~45 years old, Healthy Adult Male Subject
* Body Weight ≥ 50kg and Ideal Body Weight ≤ ±20%

Exclusion Criteria:

* ALT or AST > 1.25 times (Upper Normal Range)
* Total Bilirubin > 1.5 times (Upper Normal Range)
* CPK > 2 times (Upper Normal Range)
* BUN or Creatinine > Normal Range
* Systolic BP > 160mmHg or < 80mmHg, Diastolic BP > 100mmHg or < 50mmHg

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Cmax,ss | 48h
  Pharmacokinetic of Oxycodone
AUCτ | 24h
  Pharmacokinetic of Oxycodone

SECONDARY OUTCOMES:
Tmax | 48h
  Pharmacokinetic of Oxycodone
t1/2 | 48h
  Pharmacokinetic of Oxycodone
Vz/f | 48h
  Pharmacokinetic of Oxycodone
CL/F | 48h
  Pharmacokinetic of Oxycodone
Cmin,ss | 48h
  Pharmacokinetic of Oxycodone
Cave,ss | 48h
  Pharmacokinetic of Oxycodone
degree og fluctuation | 48h
  Pharmacokinetic of Oxycodone
  (Cmax,ss-Cmin,ss)/Cave,ss
swing | 48h
  Pharmacokinetic of Oxycodone
  (Cmax,ss-Cmin,ss)/Cmin,ss
R | 48h
  Pharmacokinetic of Oxycodone
  Accumulation index

CONTACTS AND LOCATIONS:
Overall Officials: Doo-Yeoun Cho, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- AJOU University Hospital, Suwon, Gyeonggido, South Korea